CLINICAL TRIAL: NCT05236231
Title: A Single-center, Open-label, Single-dose, Randomized, 3-way Crossover Phase 1 Study in Healthy Adult Participants to Assess the Bioequivalence of the Combination of Macitentan/Tadalafil (10 mg/20 mg) Administered as a Fixed Dose Combination Formulation Compared to the Reference Free Combination of 10 mg Macitentan (Opsumit®) and 20 mg Tadalafil (Adcirca®) as Well as the Food Effect of the Fixed-dose Combination Formulation
Brief Title: A Study of Fixed Dose Combination of Macitentan/Tadalafil (10 mg/20 mg) Compared to the Reference Free Combination of Macitentan and Tadalafil in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109140; 67896062PAH1002 (Other: Actelion)
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — macitentan; Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Sequence ABC (Experimental): Participants will receive single oral dose of fixed dose combination (FDC) of macitentan/tadalafil under fasting conditions in (test) (Treatment A) Treatment Period 1 followed by single oral dose of FDC of macitentan/tadalafil under fed conditions (test) (Treatment B) in Treatment Period 2 and then single oral dose of macitentan/tadalafil under fasting conditions (reference) (Treatment C) in Treatment Period 3 on Day 1 of each Treatment Period. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC
- Treatment Sequence BCA (Experimental): Participants will receive Treatment B in Treatment Period 1 followed by Treatment C in Treatment Period 2 and Treatment A in Treatment Period 3. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC
- Treatment Sequence CAB (Experimental): Participants will receive Treatment C in Treatment Period 1 followed by Treatment A in Treatment Period 2 and Treatment B in Treatment Period 3. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC
- Treatment Sequence ACB (Experimental): Participants will receive Treatment A in Treatment Period 1 followed by Treatment C in Treatment Period 2 and Treatment B in Treatment Period 3. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC
- Treatment Sequence CBA (Experimental): Participants will receive Treatment C in Treatment Period 1 followed by Treatment B in Treatment Period 2 and Treatment A in Treatment Period 3. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC
- Treatment Sequence BAC (Experimental): Participants will receive Treatment B in Treatment Period 1 followed by Treatment A in Treatment Period 2 and Treatment C in Treatment Period 3. There will be a wash-out period of at least 12 days between Day 1 of subsequent treatment period.
  Interventions: Drug: Macitentan 10 mg; Drug: Tadalafil 20 mg; Drug: Macitentan 10 mg/Tadalafil 20mg FDC

INTERVENTIONS:
Drug: Macitentan 10 mg — Macitentan 10mg tablet will be administered orally as per assigned treatment sequence.
  Other Names: Opsumit; JNJ-67896062
Drug: Tadalafil 20 mg — Tadalafil 20mg tablet will be administered orally as per assigned treatment sequence.
  Other Names: Adcirca; JNJ-10291697
Drug: Macitentan 10 mg/Tadalafil 20mg FDC — FDC of Macitentan 10 mg/Tadalafil 20 mg will be administered orally as single dose tablets.
  Other Names: ACT-064992D

SUMMARY:
The purpose of this study is to demonstrate bioequivalence on the primary pharmacokinetic (PK) parameters between macitentan and tadalafil administered as a fixed dose combination (FDC) (test) of macitentan/tadalafil and the co- administered free combination (reference) of macitentan (Opsumit) and tadalafil (Adcirca) in fasted conditions in healthy adult participants; and to evaluate the effect of food on the primary PK parameters of macitentan and tadalafil administered as an FDC of macitentan/tadalafil in fed versus fasted conditions in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination and medical history, performed at screening. If there are any abnormalities, they must be considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Systolic blood pressure (SBP) between 100 and 145 millimeters of mercury (mm Hg) (inclusive), diastolic blood pressure (DBP) between 50 and 90 mm Hg (inclusive), and pulse rate between 45 and 90 beats per minute (inclusive) at screening, supine for at least 5 minutes and after 3 minutes of standing
* Twelve-lead electrocardiogram (ECG) without clinically relevant abnormalities, at the discretion of the investigator, measured after the participant is supine for at least 5 minutes, at screening
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after the last study intervention intake
* Willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to macitentan, tadalafil, or drug of the same class, or its excipients
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study intervention(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Veins unsuitable for intravenous puncture on either arm (example, veins that are difficult to locate, access, or puncture, and veins with a tendency to rupture during or after puncture)
* Known hereditary degenerative retinal disorders, including retinitis pigmentosa

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Macitentan and its Metabolite JNJ-68212820, and Tadalafil. | Predose up to 216 hours (up to Day 10)
  Cmax is defined as the maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration Time Curve of Macitentan, its Metabolite JNJ-68212820, and Tadalafil from Time Zero to Time of the Last Quantifiable Concentration (AUC [0-Last]) | Predose up to 216 hours (up to Day 10)
  AUC (0-last) is defined as area under the plasma analyte concentration time curve of macitentan, its metabolite JNJ-68212820 and tadalafil from time 0 to the time of the last quantifiable (non-below quantification limit [non-BQL]) concentrations.
Area Under the Plasma Concentration Time Curve of Macitentan and its Metabolite JNJ-68212820, and Tadalafil from Time Zero to Infinite time (AUC [0-Infinity]) | Predose up to 216 hours (up to Day 10)
  AUC (0-infinity) is defined as area under the plasma concentration-time curve of macitentan and its metabolite JNJ-68212820, and tadalafil from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z) where C(last) is the last observed measurable (non-BQL) plasma analyte concentration.

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Analyte Concentration (Tmax) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  Tmax is defined as actual sampling time to reach the maximum observed plasma analyte concentration.
Area Under the Plasma Concentration Versus Time Curve of Macitentan and its Metabolite JNJ-68212820, Tadalafil From Time Zero up to 72 Hours Post Dosing (AUC72h) | Predose up to 216 hours (up to Day 10)
  (AUC 0-72h) is defined as the area under the plasma concentration-time curve of macitentan and its metabolite JNJ-68212820, tadalafil from time 0 to 72 hours postdose, calculated by linear-linear trapezoidal summation.
Apparent Elimination Half-Life (t1/2) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  t1/2 is defined as apparent elimination half-life calculated as 0.693/lambda(z).
Apparent Terminal Elimination Rate Constant (lambda z) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  Apparent terminal elimination rate constant is estimated by linear regression using the terminal log-linear phase of the log-transformed concentration versus time curve.
Total Apparent Oral Clearance (CL/F) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  CL/F is defined as total apparent oral clearance calculated as dose/AUC(0-infinity).
Apparent Volume of Distribution (Vd/F) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  Vd/F is defined as apparent volume of distribution calculated as dose/(lambda(z) *AUC (0 to infinity).
Last Observed Measurable Plasma Concentration (Clast) of Macitentan and its Metabolite JNJ-68212820, Tadalafil | Predose up to 216 hours (up to Day 10)
  Clast is defined as the last observed measurable (non-BQL) plasma concentration of macitentan and its metabolite JNJ-68212820, Tadalafil.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (1):
- PRAHS, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency